CLINICAL TRIAL: NCT02309905
Title: Evaluation of Tele-expertise for Inmates With a Dermatological Lesion
Acronym: TLM-Inmates
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: Teledermatology for Inmates
Record Dates: First submitted 2014-11-27; First posted 2014-12-05 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-12

CONDITIONS: Skin Disease
Keywords: inmates; skin lesion; telemedicine
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control group before telemedicine: Inmates of prisons not having telemedicine before implementation of telemedicine in prisons having telemedicine
- Control group after telemedicine: Inmates of prisons not having telemedicine after implementation of telemedicine in prisons having telemedicine
- Exposed group, before telemedicine: Inmates of prisons having telemedicine before implementation of telemedicine
- Exposed group, after telemedicine: Inmates of prisons having telemedicine after implementation of telemedicine
  Interventions: Device: Telemedicine

INTERVENTIONS:
Device: Telemedicine — Inmates of prisons having telemedicine after implementation of telemedicine
  Groups: Exposed group, after telemedicine

SUMMARY:
The purpose of this study is to determine whether Tele-expertise would be effective and cost-effective by reducing the number of secure transportations for inmates in need of a dermatological consultation

ELIGIBILITY:
Inclusion Criteria:

* Dermatological expertise required

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inmates
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of a dermatological expertise among those required | 1 month after the end of the study

SECONDARY OUTCOMES:
Number of hospitalizations for a dermatological reason | 1 month after the end of the study
Overall costs | 6 months after the end of the study
Time to a dermatological expertise | 1 month after the end of the study
Number of usual consultations needed after Tele-expertise | 1 month after the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: François Moreau, MD, Principal Investigator — Versailles Hospital; Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - UCSA Osny, Cergy-Pontoise
  - UCSA Meaux, Meaux
  - UCSA Nanterre, Nanterre
  - UCSA Réau, Réau
  - UCSA Villepinte, Villepinte

REFERENCES:
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736
- [Derived] Zarca K, Charrier N, Mahe E, Guibal F, Carton B, Moreau F, Durand-Zaleski I. Tele-expertise for diagnosis of skin lesions is cost-effective in a prison setting: A retrospective cohort study of 450 patients. PLoS One. 2018 Sep 24;13(9):e0204545. doi: 10.1371/journal.pone.0204545. eCollection 2018. PMID 30248151
- [Derived] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558